CLINICAL TRIAL: NCT04678622
Title: Proof of Concept: Clinical Validation Study of Personalized Orthopedic Splints With 3D Technology in Patients With Rhizarthrosis
Brief Title: Clinical Validation Study of Personalized Orthopedic Splints With 3D Technology in Patients With Rhizarthrosis
Status: Completed | Type: Observational
Sponsor: Optimus3D S.L. (Industry)
Collaborators: Biobizkaia Health Research Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: BIOFERULA3D
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis of the Small Joints of the Hand
Keywords: Orthotic Devices; Biosplint 3D; Rhizarthrosis; Eaton-Littler I / II clasification; 3D technology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Classic Orthrosis: Group of patients who they will wear the usual splint indicated by the servicio physicians
- 3D Orthrosis: Group of patients who they will wear the personalized splint designed by the company OPTIMUS 3D.
  Interventions: Device: Bioferula3D

INTERVENTIONS:
Device: Bioferula3D — Custom splint with 3D technology classified as a custom medical device
  Groups: 3D Orthrosis

SUMMARY:
Osteoarthritis of the hand is a chronic joint disease that usually affects one or more of the finger joints and it is a major cause of disability. Radiology and the Eaton-Littler classification (Stages I-II-III-IV) are used for its diagnosis. The treatment of stages I, II and in some cases of stage III, is based on pharmacological and rehabilitation measures, including the use of orthoses or splints.

The development of Biosplint 3D will allow a qualitative leap forward in the search for an intelligent solution for patients with rhizarthrosis (Degenerative alteration of the trapezius-metacarpal joint (TMJ) characterized by a progressive deterioration of the articular surfaces and new bone formation in them).

The aim of the study is to assess the feasibility of applying a personalized splint versus a conventional one. It is not a design aimed at evaluating the efficacy of such treatment. It is a prospective study with two arms, open with 1:1 allocation.

The study includes a recruitment visit and two follow-up visits, one at a month and a final visit at 3 months. Patients with a new diagnosis of osteoarthritis of the trapeziometacarpal joint are included. One group of patients wears the usual splint indicated by the personalized doctors of the Service and the other group wears the 3D bi-splint.

The main variable is pain, which will be measured by a visual analog scale (VAS). In addition, the DASH questionnaire (Disabilities of the Arm, Shoulder and Hand) and questions about patient satisfaction with the use of splints will be used.

DETAILED DESCRIPTION:
Osteoarthritis of the TMJ is a disease present in a large part of the general population. The symptomatic prevalence is estimated at 6-8% of the population, although its radiological prevalence would be 29-76%. Its diagnosis is basically clinical, although radiological tests are very useful to confirm it and to typify the evolution of the disease.

The TMJ has a great range of mobility, since it basically serves to oppose the thumb to the rest of the fingers and to carry out grasping or pinching actions, which is why it is of great use and of great utility in everyday life. This range of movements is favored by being a not very congruent joint, but this fact also explains the tendency to instability, which can lead to abnormal movements between the joint surfaces, which ultimately lead to the development of osteoarthritis of the joint. joint. Over time, a subluxation occurs and the first metacarpal tends to approach the rest of the fingers, producing an adduction. This osteoarthritis leads to pain and functional disability. The pain is usually greater when the joint is stressed, during pincer movements.

• Conventional orthoses

Currently there are several types of splints on the market made of temperature-moldable plastic material, a splint that has multiple disadvantages in terms of manufacture:

* Polypropylene shrinks with heat, so it must be taken into account when designing. In addition, special care must be taken when heating and thermoforming it since the orthosis can collapse more easily. If it is not heated, it may not thermoform well.
* You cannot make rectifications, so you have to be careful with the mold and make screeds or modifications before adapting the polypropylene, since once it has been fused no changes can be made.

Another type of splints that exist on the market are splints made of polyethylene sheets adjustable with velcro. The disadvantage of these splints is their instability in immobilization: they do not hold firmly, since they do not fit perfectly to the affected area.

• Advantages of the 3D bioferula

The splints developed using this method have a series of advantages both in manufacturing and for patients, among which we can highlight:

* Increase the precision in the design of the splint to place it in the affected area.
* Reduce the weight of the splint in order to lead a more agile life.
* Improve perspiration.
* Water resistance, which will improve hygiene, the patient can even bathe with the splint on.
* Greater mobility. The "pincer" movement will not be affected.
* Allow air circulation.
* Improve aesthetic appearance: simple splint design that can be covered if the patient considers it so, for example, with gloves.
* Manufacturing times: the 3D model is made in 3 hours and can be in use by the patient in 72 hours.
* It can be made with fully recyclable materials.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis of the trapeziometacarpal joint.
* Radiological stage of Eaton-Littler classification I / II.
* Patients in whom the placement of a discharge splint is clinically indicated.
* Score between 3 and 7 on the VAS pain scale (range 0 to 10).

Exclusion Criteria:

* Previous treatment of osteoarthritis of the trapeziometacarpal joint.
* Refuses to participate in the study.
* Disabilities that prevent the completion of the questionnaires.
* Presence of severe deformations in the hand.
* Presence of other alterations, such as carpal tunnel syndrome, tendonitis or chronic inflammatory arthropathies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a new diagnosis of osteoarthritis of the trapeziometacarpal joint
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Pain measured: Change of pain in patients with clasic orthrosis compared to the orthrosis designed using 3D technology | Pain measurement by visual analog scale is performed at the baseline visit, at the second visit (one month later) and at the third follow-up visit (end of the study) which will take place at the third month of follow-up (between 11-14 weeks).
  By visual analog scale from 0 (no pain) to 10 (unbereable pain)

SECONDARY OUTCOMES:
3D orthoses change functionality | Functionality is performed at the baseline visit, at the second visit (one month after) and at the third follow-up visit (end of the study), which will take place at the third month of follow-up (between 11-14 weeks).
  By DASH (10) scale consists of 30 items. In addition, there are 2 optional modules, with 4 items each one of them, that will measure the impact of an upper limb injury when playing musical instruments and when doing sports or working. Each item is scored from 1 to 5, with increasing values depending on the intensity of the symptoms. The score of the items is added to obtain a total score, which can range between 30 and 150 points and which is transformed into a scale from 0 (best possible score) to 100 (worst possible score).
  The DASH scale makes it possible to assess the disability perceived by the patient to perform various activities, including activities of daily living and symptoms such as pain, stiffness or loss of strength.
Satisfaction and compliance are equally superior in the 3D orthosis. | Satisfaction is performed at the second visit (one month after) and at the third follow-up visit (end of the study), which will take place at the third month of follow-up (between 11-14 weeks).
  By satisfaction scale composed of 6 items (each of them scored from 0 to 10):
  1. What is your level of satisfaction with the splint?
  2. Has the splint helped decrease your pain?
  3. Has the splint helped you maintain your daily activities?
  4. Has your quality of life improved?
  5. How comfortable was the use of the splint?
  6. How easy was it to follow the instructions for using the splint?

OTHER OUTCOMES:
There are no relevant differences between the two orthoses in terms of fist force and clamp force. | It is performed at the second visit (one month after) and at the third follow-up visit (end of the study), which will take place at the third month of follow-up (between 11-14 weeks).
  By gripping force, using a dynamometer in the consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Iñigo Cearra Guezuraga, IP, Principal Investigator — Biobizkaia Health Research Institute
Locations (2):
- Spain (2):
  - Optimus 3D S.L., Vitoria-Gasteiz, Alava
  - Hospital Universitario Basurto, Bilbao, Vizcaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper C, Egger P, Coggon D, Hart DJ, Masud T, Cicuttini F, Doyle DV, Spector TD. Generalized osteoarthritis in women: pattern of joint involvement and approaches to definition for epidemiological studies. J Rheumatol. 1996 Nov;23(11):1938-42. PMID 8923371
- [Background] Gomes Carreira AC, Jones A, Natour J. Assessment of the effectiveness of a functional splint for osteoarthritis of the trapeziometacarpal joint on the dominant hand: a randomized controlled study. J Rehabil Med. 2010 May;42(5):469-74. doi: 10.2340/16501977-0542. PMID 20544159
- [Background] Hirschfeld M, Galan A, Arenas J, Del Aguila B, Benitez-Parejo N, Costa JA, Guerado E. [Inter-observer agreement on the Eaton-Littler classification of trapeziometacarpal joint osteoarthritis]. Rev Esp Cir Ortop Traumatol. 2014 Jul-Aug;58(4):237-41. doi: 10.1016/j.recot.2014.01.006. Epub 2014 May 10. Spanish. PMID 24821479
- [Background] Eaton RG, Littler JW. Ligament reconstruction for the painful thumb carpometacarpal joint. J Bone Joint Surg Am. 1973 Dec;55(8):1655-66. No abstract available. PMID 4804988
- [Background] Spaans AJ, van Minnen LP, Kon M, Schuurman AH, Schreuders AR, Vermeulen GM. Conservative treatment of thumb base osteoarthritis: a systematic review. J Hand Surg Am. 2015 Jan;40(1):16-21.e1-6. doi: 10.1016/j.jhsa.2014.08.047. PMID 25534834
- [Background] Barron OA, Glickel SZ, Eaton RG. Basal joint arthritis of the thumb. J Am Acad Orthop Surg. 2000 Sep-Oct;8(5):314-23. doi: 10.5435/00124635-200009000-00005. PMID 11029559
- [Background] Bani MA, Arazpour M, Kashani RV, Mousavi ME, Maleki M, Hutchins SW. The effect of custom-made splints in patients with the first carpometacarpal joint osteoarthritis. Prosthet Orthot Int. 2013 Apr;37(2):139-44. doi: 10.1177/0309364612454047. Epub 2012 Aug 22. PMID 22918521
- [Background] Hamann N, Heidemann J, Heinrich K, Wu H, Bleuel J, Gonska C, Bruggemann GP. Stabilization effectiveness and functionality of different thumb orthoses in female patients with first carpometacarpal joint osteoarthritis. Clin Biomech (Bristol). 2014 Dec;29(10):1170-6. doi: 10.1016/j.clinbiomech.2014.09.007. Epub 2014 Sep 19. PMID 25266241
- [Background] Chiu NF, Huang TY, Kuo CC, Lin CW, Lee JH. Organic-based plasmonic emitters for sensing applications. Appl Opt. 2013 Mar 1;52(7):1383-8. doi: 10.1364/AO.52.001383. PMID 23458789

DOCUMENTS (2):
  • Study Protocol (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT04678622/Prot_000.pdf
  • Informed Consent Form (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT04678622/ICF_001.pdf